CLINICAL TRIAL: NCT04310891
Title: Validation of Markerless Image Guidance Using Intrafraction Kolovoltage X-ray Imaging Using Implanted Fiducials: Phase I Observational Study of Lung Cancer Radiotherapy
Brief Title: Markerless Image Guidance Using Intrafraction Kolovoltage X-ray Imaging for Lung Cancer Radiotherapy
Acronym: VALKIM
Status: Active, not recruiting | Type: Observational
Sponsor: Royal North Shore Hospital (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Dasantha Jayamanne, Radiation Oncologist, Royal North Shore Hospital
Other Study IDs: VALKIM
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Markerless Image Guidance; Intrafraction Kolovoltage X-ray Imaging
Keywords: Lung Cancer; Radiotherapy; Fiducials; Markerless Tumour Tracking
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Markerless: Markerless Tumour Tracking will be used to observe the radiation beam is accurately targeting the tumour.
  Interventions: Radiation: Markerless Tumour Tracking

INTERVENTIONS:
Radiation: Markerless Tumour Tracking — Intrafraction Kolovoltage X-ray Imaging using Fiducials

SUMMARY:
In radiotherapy, tumour tracking allows us to ensure the radiation beam is accurately targeting the tumour while it moves in a complex and unpredictable way. Most tumour tracking techniques require the implantation of fiducial markers around the tumour. Markerless Tumour Tracking negates the need for implanted markers, enabling accurate and optimal cancer radiotherapy in a non-invasive way.

DETAILED DESCRIPTION:
We will perform a phase I observational trial investigating the feasibility of the Markerless Tumour Tracking technology. Markerless Tumour Tracking will be integrated with existing treatment machines to provide real-time monitoring of tumour motion during treatment delivery. Eligible patients are implanted with fiducial markers, which act as the ground truth for evaluating the accuracy of Markerless Tumour Tracking. The patients will undergo the current standard of care radiotherapy, with the exception that kilovoltage x-ray images will be acquired continuously during treatment delivery and used to calculate online Markerless Tumour Tracking. Markerless Tumour Tracking determines the mean tumour position calculated over the most recent 15 seconds and displays shifts exceeding 3 mm.

The trial will be a single-institution study recruiting only at RNSH Radiation Oncology Department.

As this trial investigates feasibility, our focus will be on estimating the proportion of treatment time in which the Markerless Tumour Tracking is within acceptable limits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older.
2. Has provided written Informed Consent for participation in this trial and is willing to comply with the study.
3. Patients undergoing external beam radiotherapy.
4. Histologically proven Stage I NSCLC or oligometastatic lung metastases (3 or less).
5. Diagnostic CT prior to insertion of fiducial markers.
6. Patient must be able to have fiducial markers placed in the lung (if on anticoagulants, must be cleared by LMO or cardiologist).
7. ECOG performance status 0-2.
8. A maximum of three metastases to the lung from any non-haematological malignancy. Multiple metastases will be treated separately.
9. 1 cm ≤ Tumour diameter in any dimension ≤ = 5 cm.
10. The distance between the tumour centroid and the top end of the diaphragm is <=8 cm.

Exclusion Criteria:

1. Patient has low respiratory performance as evaluated by the physicians.
2. Previous high-dose thoracic radiotherapy.
3. Less than one fiducial marker implanted in the lung.
4. Fiducial markers are too far from the tumour centroid (>9 cm).
5. Cytotoxic chemotherapy within 3 weeks of commencement of treatment, or concurrently with treatment. Hormonal manipulation agents are allowable (e.g. aromatase inhibitors, selective oestrogen receptor modulators, and gonadotropin releasing hormone receptor modulators).
6. Targeted agents (such as sunitinib, bevacizumab and tarceva) within 7 days of commencement of treatment, concurrently with treatment or 7 days after radiotherapy.
7. Women who are pregnant or lactating.
8. Unwilling or unable to give informed consent.
9. Unwilling or unable to complete quality of life questionnaires.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults >=18 years with NSCLC
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Markerless Tumour Tracking | 6 months after recruitment
  to demonstrate the feasibility of Markerless Tumour Tracking for motion-adaptive lung cancer radiotherapy as assessed by agreement between markerless and marker-based tracking within 3 mm for at least 80% of the beam-on time as assessed in off-line analyses.

SECONDARY OUTCOMES:
Markerless Tumour Tracking outcome | 6 months after treatment of last fraction
  To identify cohort of patients on which markerless Tumour tracking performs well or poorly
Accuracy | 6 months after treatment of last fraction
  To quantify the accuracy of marker-based tracking by comparison with MV-kV triangulation or visual inspection
Magnitude | 6 months after treatment of last fraction
  To investigate the magnitude of surrogacy of lung tumour motion, ie the difference between tumour motion and implanted marker motion
Correlation | 6 months after treatment of last fraction
  To investigate the correlation between external and internal motion using infrared/optical imaging
Suitability | 6 months after treatment of last fraction
  To investigate the suitability and frequency of correcting for tumour baseline shifts based on a variety of tolerance criteria and with different methods
Frequency | 6 months after treatment of last fraction
  To investigate the frequency of correcting for tumour baseline shifts based on a variety of tolerance criteria and with different methods
Feasibility of outcomes prediction | 6 months after treatment of last fraction
  To investigate the feasibility of predicting treatment outcomes based on patient and imaging information
Outcomes | 6 months after treatment of last fraction
  Participants will be followed for 2 years to determine patient outcomes, including radiation therapy toxicity, local control (whether the tumour has spread) and survival
Historical | 6 months after treatment of last fraction
  2 year outcomes will be compared to historical outcomes reported from our lung Departmental SBRT database
Ineligibility | 6 months after treatment of last fraction
  To record the number of patients ineligible after marker insertion due to positioning of markers, or due to complications with the implantation procedure
Radiomic Features | 6 months after treatment of last fraction
  To investigate the feasibility of extracting radiomic features from CT, CBCT, and kV images to predict tumour volumes, tracking accuracy, treatment response, and patient outcomes.
X-ray dose | 6 months after treatment of last fraction
  To report additional x-ray dose caused by imaging during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dasantha Jayamanne, MD, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, Saint Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided